CLINICAL TRIAL: NCT07154121
Title: Efficacy Evaluation of 5-Fluorouracil as an Adjuvant to Endoscopic Dacryocystorhinostomy in Managing Primary Acquired Nasolacrimal Duct Obstruction With Small Lacrimal Sac: A Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025KYPJ065
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Primary Acquired Nasolacrimal Duct Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: 5-fluorouracil group
- control group (Active Comparator)
  Interventions: Other: saline group

INTERVENTIONS:
Drug: 5-fluorouracil group — Patients in the intervention group underwent standard En-DCR surgery, with all procedures performed by the same senior oculoplastic surgeon; After suturing to create a new nasolacrimal duct during surgery, Schirmer strips were placed at the ostium to measure its size and photographed for record-keeping. The ostium was then covered with a gelatin sponge soaked in 12.5 mg/mL 5-fluorouracil for 3 minutes, after which the gelatin sponge was removed and the area thoroughly rinsed with saline.
  Arms: experimental group
Other: saline group — Patients in the intervention group underwent standard En-DCR surgery, with all procedures performed by the same senior oculoplastic surgeon; Similarly, after suturing to create a new nasolacrimal duct during surgery, Schirmer strips were placed at the ostium to measure its size and photographed for record-keeping. The ostium was then covered with a gelatin sponge soaked in saline solution for 3 minutes, after which the gelatin sponge was removed and the ostium was thoroughly rinsed with saline solution.
  Arms: control group

SUMMARY:
Primary acquired nasolacrimal duct obstruction (PANDO) is a lacrimal duct obstruction disease characterized by inflammatory fibrosis of the nasolacrimal duct, with primary symptoms including epiphora and increased secretions, commonly seen in middle-aged and elderly women over 40 years of age . The pathogenesis of PANDO remains unclear, and there are no effective pharmacological treatments. Dacryocystorhinostomy (DCR) is currently considered the primary treatment for PANDO, as it restores tear drainage by creating an alternative drainage pathway between the lacrimal sac and the nasal cavity.

The surgical techniques for DCR primarily include external DCR (Ex-DCR) and endoscopic DCR (En-DCR), with En-DCR first proposed by McDonogh and Meiring in 1989. In recent years, with the advancement of endoscopic sinus surgery techniques, En-DCR has gained widespread recognition in the treatment of PANDO, as it not only minimizes surgical trauma and accelerates postoperative recovery but also leaves no external scars. In recent years, with the advancement of endoscopic surgical techniques, En-DCR has gained widespread recognition in the treatment of PANDO, as it not only causes minimal surgical trauma and facilitates rapid postoperative recovery; but also leaves no external scars, making it more aesthetically pleasing; and can simultaneously correct nasal cavity abnormalities such as deviated nasal septum and sinusitis. Recent studies indicate that the surgical success rate of En-DCR can reach 84%-94%, comparable to traditional external surgery Recent studies have shown that the surgical success rate of En-DCR can reach 84%-94%, comparable to traditional external approaches.

Although the prognostic factors associated with En-DCR outcomes have not yet been fully elucidated, it has been demonstrated that lacrimal sac size is one of the key indicators for predicting the efficacy of En-DCR surgery, and a small lacrimal sac is a major risk factor for En-DCR surgical failure. In patients with normal-sized lacrimal sacs, creating a larger bone window can better expose the lacrimal sac, thereby forming a larger lacrimal sac flap, making the lacrimal sac opening wider, and reducing the risk of postoperative obstruction. However, in patients with small lacrimal sacs, even if the bone window is intentionally enlarged during surgery, the resulting lacrimal sac flap remains small due to the inherent small size of the lacrimal sac, making it difficult to achieve proper alignment with the nasal mucosal flap at the anterior margin of the hook process, resulting in poor anastomotic outcomes. In PANDO cases, the primary cause of surgical failure is often related to abnormal healing of the anastomotic site postoperatively, particularly scar formation at the surgical site and scar-induced closure of the bone window. Compared to patients with normal-sized lacrimal sacs, patients with small lacrimal sacs are more prone to osteotomy site closure due to granulation tissue proliferation postoperatively, thereby reducing surgical successrates. Therefore, preventing fibrous proliferation at the osteotomy site may be key to improving the success rate of En-DCR treatment for small lacrimal sac-type PANDO.

Antimetabolite drugs are frequently used to treat various ocular lesions characterized by non-tumor cell proliferation. 5-Fluorouracil (5-FU) is one such drug, which inhibits DNA synthesis by blocking thymidine kinase, an enzyme involved in collagen gene expression. In vitro studies have shown that 5-FU interferes with the biosynthesis of F-actin and prevents fibroblast migration; 5-FU can inhibit scar formation by suppressing fibroblast proliferation; and 5-FU can prolong wound healing time. 5-FU is now widely used to inhibit fibroblast proliferation and scar formation within the filter after glaucoma filtration surgery, demonstrating good safety and efficacy. This study is the first to explore the efficacy of 5-fluorouracil as an adjunct to En-DCR therapy for small lacrimal sac PANDO, aiming to provide a new adjunctive treatment strategy for patients with small lacrimal sac PANDO.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with small lacrimal sac-type PANDO based on clinical symptoms, lacrimal duct irrigation, and CT lacrimal duct angiography (minimum diameter on lacrimal sac angiography ≤3 mm);
2. Patients aged 18 years or older;
3. Patients with no history of drug allergies (including 5-FU, contrast agents, or other substances that may affect participation in this study);
4. Patients who have provided informed consent and signed the informed consent form.

Exclusion Criteria:

1. Previously underwent nasolacrimal duct surgery;
2. Nasolacrimal duct obstruction secondary to facial surgery, sinus disease, tumors, trauma, or revision DCR;
3. Severe sinusitis or deviated nasal septum;
4. Acute dacryocystitis;
5. Patients with chronic debilitating conditions such as diabetes, malignant tumors, or malnutrition;
6. Patients with systemic diseases such as sarcoidosis or Wegener's granulomatosis that may promote scar formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate in patients with small lacrimal sac type PANDO at six months post-En-DCR surgery | Six months after surgery
  Surgical success is defined as: the patient is asymptomatic/has improved symptoms and has a FICI score of ≥3 on endoscopic examination.

SECONDARY OUTCOMES:
Surgical success rates for small lacrimal sac type PANDO patients at three weeks and three months post-En-DCR surgery | three weeks and three months after surgery
  Surgical success is defined as: the patient is asymptomatic/has improved symptoms and has a FICI score of ≥3 on endoscopic examination.
Changes in stoma size three months after surgery | three months after surgery
  Both groups of stomas formed during surgery were measured using Schirmer strips as a reference, and images were captured. The size of the stomas was measured using ImageJ software. The sizes of the stomas measured during follow-up were compared with the initial sizes of the stomas formed during surgery.
Incidence of complications during treatment | Six months after surgery
  Observe whether patients experience complications such as abnormal epistaxis, mucosal necrosis, mucosal atrophy, wound infection, or delayed wound healing after the stoma is soaked with the antimetabolite drug 5-FU during surgery. Simultaneously assess whether the drug has any adverse effects on the patient's cornea, conjunctiva, and overall condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No